CLINICAL TRIAL: NCT06118489
Title: Evaluation of the Effects of Different Anesthetic Gases on Hemodynamics, Arterial Oxygenation and Pulmonary Mechanics in Spinal Surgery.
Brief Title: Effects of Different Anesthetic Gases on Hemodynamics, Arterial Oxygenation and Pulmonary Mechanics
Status: Completed | Type: Observational
Sponsor: Sultan Abdulhamid Han Training and Research Hospital, Istanbul, Turkey (Other)
Responsible Party: Principal Investigator, Yadigar Yılmaz, principal investigator, Sultan Abdulhamid Han Training and Research Hospital, Istanbul, Turkey
Other Study IDs: HamidiyeKAEK-98172
Record Dates: First submitted 2023-10-31; First posted 2023-11-07 (Actual); Last update posted 2025-06-10 (Actual); Status verified 2025-06

CONDITIONS: Oxygenation; Spinal Surgery; Sevoflurane; Desflurane

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (2):
- sevoflurane
- desflurane

SUMMARY:
The bronchodilator effects of volatile anesthetics have been the subject of many clinical studies. It is known that all volatile anesthetics, especially halothane, have similar effects. Sevoflurane has been shown to reduce airway resistance more than halothane and isoflurane. Desflurane is difficult to use as an induction agent due to its harsh and extremely pungent odor and airway irritating effect. However, it has been shown that the risk of cough, respiratory arrest and laryngospasm is no different from sevoflurane when administered after intravenous induction. Although it irritates the airway, it is thought to have a bronchodilation effect as it stimulates the sympathetic system.

In spinal surgeries, prone position is required to access the operating field. When the patient is placed in the prone position, pulmonary physiology are affected. In the prone position, V/Q mismatch decreases and arterial oxygenation increases. However, lung compliance decreases and the peak inspiratory pressure required to reach the required tidal volume increases. The main purpose of this study is the effect of volatile agents on lung mechanics and oxygenisation in the prone position.

ELIGIBILITY:
Inclusion Criteria:

* 18-65 years old
* ASA1-2
* Patients planned to undergo spinal surgery

Exclusion Criteria:

* 1 - Lung disease
* BMI 35 and above
* Smokers
* Those under the age of 18 and over the age of 65
* Hepatorenal disease
* Reynaud's disease
* Burger disease
* Hypotensive patient
* Neuromuscular disease
* Those who have had thoracic surgery before
* Those with bad Allen test results

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: ASA 1-2 patients between the ages of 18 and 65 who are scheduled for spinal surgery will be included in the study.
Sampling Method: Probability Sample
Enrollment: 50 (Actual)
Dates: Start 2023-12-01 (Actual); Primary Completion 2024-02-01 (Actual); Study Completion 2024-02-01 (Actual)

PRIMARY OUTCOMES:
compliance | 2 hour
  pulmonary compliance before, during and after prone position

CONTACTS AND LOCATIONS:
Locations (1):
- Yadigar Yılmaz, Istanbul, Turkey (Türkiye)